CLINICAL TRIAL: NCT03017326
Title: Paediatric Hepatic International Tumour Trial
Acronym: PHITT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Fundació Institut Germans Trias i Pujol (Other); University Hospital Munich (Other); University Hospital, Bonn (Other); University of Kiel (Other); University Hospital Tuebingen (Other); University of Padova (Other); Ludwig-Maximilians - University of Munich (Other); Medical University of Gdansk (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other); Motol University Hospital (Other); Rennes University Hospital (Other); Children's University Hospital, Ireland (Other); University of Oslo (Other); Princess Maxima Center for Pediatric Oncology (Other); Andaluz Health Service (Other Government); Swiss Pediatric Oncology Group (Other); Gothia Forum - Center for Clinical Trial (Other); The Leeds Teaching Hospitals NHS Trust (Other); Bambino Gesù Hospital and Research Institute (Other); Newcastle University Centre for Cancer, Newcastle (Unknown); Experimental Cancer Medicine Centres (Other); XenTech, Evry (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: RG_15-114
Record Dates: First submitted 2016-12-14; First posted 2017-01-11 (Estimated); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Hepatoblastoma; Carcinoma, Hepatocellular
MeSH Terms: conditions — Hepatoblastoma; Carcinoma, Hepatocellular | interventions — Cisplatin; Doxorubicin; Carboplatin; Fluorouracil; Vincristine; Etoposide; Irinotecan; Gemcitabine; Oxaliplatin; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group A Very Low Risk HB (Other): Patients with well differentiated foetal histology will receive 2 cycles of Cisplatin (2x 100mg/m2). Patients will non-well differentiated histology will be followed up only (no intervention).
  Interventions: Drug: Cisplatin
- Group B Low Risk HB (Active Comparator): Patients who are resected after 2 cycles of Cisplatin will be randomised to receive 4 or 6 cycles of Cisplatin overall (80mg/m2). Patients who are not resected will continue to receive up to 6 cycles of Cisplatin (80mg/m2) until resection.
  Interventions: Drug: Cisplatin
- Group C Intermediate Risk HB (Active Comparator): Patients will be randomised to receive Cisplatin (80mg/m2), Carboplatin (500mg/m2) and Doxorubicin (60mg/m2) as SIOPEL-3HR (5 cycles), Cisplatin (100mg/m2), Doxorubicin (60mg/m2) 5-Fluorouracil (600mg/m2) and Vincristine (4.5mg/m2) as C5VD (6 cycles), or 6 cycles of high dose Cisplatin (100mg/m2)
  Interventions: Drug: Cisplatin; Drug: Doxorubicin; Drug: Carboplatin; Drug: 5Fluorouracil; Drug: Vincristine
- Group D High Risk HB (Active Comparator): Patients will receive SIOPEL-4 regimen (Cisplatin 70mg/m2, Doxorubicin 30mg/m2) then have surgery. Post surgery, patients with remaining metastases will be randomised to receive 6 cycles of either Carboplatin (500mg/m2) and Doxorubicin (40mg/m2) alternating with Carboplatin (800mg/m2) and Etoposide (400mg/m2), or Carboplatin (500mg/m2) and Doxorubicin (40mg/m2) alternating with Vincristine (3mg/m2) and Irinotecan (250mg/m2). Patients with no metastases will receive the standard treatment of 3 cycles of Carboplatin (500mg/m2) and Doxorubicin (40mg/m2).
  Interventions: Drug: Cisplatin; Drug: Doxorubicin; Drug: Carboplatin; Drug: Vincristine; Drug: Etoposide; Drug: Irinotecan
- Group E Resected HCC (Other): Patients with an underlying predisposition to HCC through genetic, viral or metabolic conditions will be followed up (no intervention). De novo or fibrolamellar HCC patients will receive 4 cycles of PLADO regimen (Cisplatin (80mg/m2) and Doxorubicin (60mg/m2)) over 4 cycles.
  Interventions: Drug: Cisplatin; Drug: Doxorubicin
- Group F Unresected HCC (Active Comparator): Patients will be randomised to receive up to 6 cycles of PLADO (Cisplatin 80mg/m2, Doxorubicin 60mg/m2) with Sorafenib (300mg/m2) or up to 8 cycles of PLADO with Sorafenib and GEMOX (Gemcitabine 1000mg/m2, Oxaliplatin 100mg/m2) with Sorafenib (300mg/m2)
  Interventions: Drug: Cisplatin; Drug: Doxorubicin; Drug: Gemcitabine; Drug: Oxaliplatin; Drug: Sorafenib

INTERVENTIONS:
Drug: Cisplatin — Arms A and B - cisplatin is used alone Arms C, D, E and F - cisplatin us used in combination
Drug: Doxorubicin — Arms C, D and E used in combination
  Arms: Group C Intermediate Risk HB; Group D High Risk HB; Group E Resected HCC; Group F Unresected HCC
Drug: Carboplatin — Arms C and D used in combination
  Arms: Group C Intermediate Risk HB; Group D High Risk HB
Drug: 5Fluorouracil — Arm C used alone
  Arms: Group C Intermediate Risk HB
Drug: Vincristine — Arms C and D used in combination
  Arms: Group C Intermediate Risk HB; Group D High Risk HB
Drug: Etoposide — Arm D used in combination
  Arms: Group D High Risk HB
Drug: Irinotecan — Arm D used in combination
  Arms: Group D High Risk HB
Drug: Gemcitabine — Arm F used in combination
  Arms: Group F Unresected HCC
Drug: Oxaliplatin — Arm F used in combination
  Arms: Group F Unresected HCC
Drug: Sorafenib — Arm used in combination
  Arms: Group F Unresected HCC

SUMMARY:
The PHITT trial is an over-arching study for patients with Hepatoblastoma (HB) and Hepatocellular Carcinoma (HCC). This trial will use a risk-adapted approach to the treatment of children diagnosed with HB.

Children with HCC will be included as a separate cohort.

DETAILED DESCRIPTION:
The trial will evaluate whether reducing treatment for low risk HB patients maintains their excellent event free survival (EFS) and decreases acute and long-term toxicity. Intensification of therapy with the use of novel agents will be evaluated in the high risk group. The trial will also compare three different regimens in intermediate risk HB.

Patients with HCC will be divided into groups based on whether the tumour is resectable or unresectable and/or metastatic.

Evaluation of the biology of HB and HCC, using the identification/validation of novel and already reported prognostic biomarkers as well as toxicity biomarkers is a key strand of this trial, so patients in all risk groups can be registered. The trial is also designed to optimise the collection of clinically annotated biologic specimens and establish the world's largest repository of blood and tissue samples from paediatric patients with HB and HCC.

The trial includes 4 randomised comparisons addressing therapeutic questions. For low risk HB patients, outcome with a total of 4 cycles of treatment is not inferior to those receiving a total of 6 cycles of treatment.

For intermediate risk patients, 3 regimens will be compared for outcome and toxicity.

For high risk patients, 2 post induction regimens will be compared for outcome. For resected HCC patients, the addition of GEMOX to PLADO regimen will be compared.

In addition the following will be assessed:

* To validate a new global risk stratification, defined by Children's Hepatic Tumours International Collaboration (CHIC)
* To evaluate clinically relevant factors, including the following:

  * Provide a comprehensive and highly-validated panel of diagnostic and prognostic biomarkers
  * Determine if paediatric HCC is a biologically different entity to adult HCC
  * Develop genomic and/or biomarker analysis to predict children who may have an increased risk of developing toxicity with chemotherapy.
* To establish a collection of clinically and pathologically-annotated biological samples.
* Evaluate a surgical planning tool for an impact on decision making processes in POST-TEXT III and IV HB

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of HB* and histologically defined diagnosis of HB or HCC.

  *Histological confirmation of HB is required except in emergency situations where:
  * a) the patient meets all other eligibility criteria, but is too ill to undergo a biopsy safely, the patient may be enrolled without a biopsy.
  * b) there is anatomic or mechanical compromise of critical organ function by tumour (e.g., respiratory distress/failure, abdominal compartment syndrome, urinary obstruction, etc.)
  * c) Uncorrectable coagulopathy
* Age ≤30 years
* Written informed consent for trial entry

Exclusion Criteria:

* Any previous chemotherapy or currently receiving anti-cancer agents
* Recurrent disease
* Previously received a solid organ transplant; other than orthotopic liver transplantation (OLT).
* Uncontrolled infection
* Unable to follow or comply with the protocol for any reason
* Second malignancy
* Pregnant or breastfeeding women

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 450 (Estimated)
Dates: Start 2017-08-24 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | From date of randomisation (or registration into the trial for non-randomised patients), until date of first failure event, assessed up to 6 years.
  Event-free survival (EFS) is defined as the time from randomisation (or registration into the trial for non-randomised patients) to first failure event. Patients who have not had an event will be censored at their last follow-up date.
  Failure events are:
  * progression of existing disease or occurrence of disease at new sites,
  * death from any cause prior to disease progression,
  * diagnosis of a second malignant neoplasm.
Response in HCC is defined as complete (CR) or partial (PR) response according to RECIST version 1.1 criteria | From date of screening assessment until date of first response assessment, up to 63 days in Group F
  Response in HCC is defined as complete (CR) or partial (PR) response according to RECIST version 1.1 criteria. The assessment will be performed after 3 cycles of PLADO, or 4 cycles of PLADO+S/GEMOX+S in Group F. Patients who are not assessable for response - e.g. because of early stopping of treatment or death - will be assumed to be non-responders.

SECONDARY OUTCOMES:
Failure-free survival (FFS) | From date of randomisation (or registration into the trial for non-randomised patients) until date of first failure event, or date of last follow up assessment, assessed up to 6 years.
  Failure-free survival (FFS) is defined as the time from randomisation (or registration into the trial for non-randomised patients) to first failure event. Patients who have not had an event will be censored at their last follow-up date.
  Failure events are:
  * progression of existing disease or occurrence of disease at new sites,
  * death from any cause prior to disease progression,
  * diagnosis of a second malignant neoplasm. failure to go to resection.
Overall survival (OS) | From date of randomisation (or registration for non-randomised patients) until date of death from any cause, or date of last follow up assessment, assessed up to 6 years.
  Overall survival (OS) is defined as the time from randomisation (or registration for non-randomised patients) to death from any cause. Patients who have not died will be censored at their last follow-up date.
Toxicity categorized and graded using Common Terminology Criteria for Adverse Events (CTCAE) | From date of start of randomised treatment until date 30 days after last treatment.
  Toxicity will be recorded in relation to each cycle of randomised treatment and will be categorized and graded using Common Terminology Criteria for Adverse Events (CTCAE)
Chemotherapy-related cardiac, nephro- and oto-toxicity using Common Terminology Criteria for Adverse Events (CTCAE) | From date of start of randomised treatment until date 30 days after last treatment.
  Chemotherapy-related cardiac, nephro- and oto-toxicity will be recorded in relation to each cycle of treatment and will be categorized and graded using Common Terminology Criteria for Adverse Events (CTCAE)
Hearing loss according to the SIOP Boston Scale | From date of registration until date of last follow up assessment, or date of death, assessed up to 6 years.
  Hearing loss will be measured according to the SIOP Boston Scale for oto-toxicity. The assessment will be performed at end of treatment (EOT) and follow up
Best Response | From date of first treatment until the date of last treatment, or until the date of first documented progression or date of death, assessed up to 6 months.
  Best Response is defined as CR or PR and is based on radiological response (RECIST v1.1) and Alpha Fetoprotein (AFP) decline. Best Response will be measured throughout treatment period. Patients who are not assessable for response - e.g. because of early stopping of treatment or death - will be assumed to be non-responders.
Surgical resectability defined as complete resection, partial resection or transplant | From date of registration until date of last follow up assessment, or date of death, assessed up to 6 years.
  Surgical resectability is defined as complete resection, partial resection or transplant
Adherence to surgical guidelines | From date of registration until date of last follow up assessment, or date of death, assessed up to 6 years.
  Adherence to surgical guidelines is defined as the local clinician's surgical decision to resect or not compared to the current SIOPEL surgical guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Madhumita Dandapani, MD PhD, Principal Investigator — University of Nottingham; Marc Ansari, MD, Principal Investigator — University of Geneva
Locations (32):
- St. Anna Kinderspital, Vienna, Austria
- Cliniques Universitaires Saint-Luc, Brussels, Woluwe-Saint-Lambert, Belgium
- University Hospital Motol, Prague, Czechia
- Kuopio University Hospital, Kuopio, Finland
- CHU de Rennes, Rennes, France
- Ludwig-Maximillians-University Munich, Munich, Germany
- Children's Health Ireland Crumlin, Dublin, Ireland
- Schneider Children's Medical Center, Petah Tikva, Israel
- Prinses Maxima Center, Utrecht, Netherlands
- Oslo University Hospital, Nydalen, Norway
- Medical University of Gdansk, Gdansk, Poland
- University Hospital Reina Sofia, Córdoba, Spain
- Hopitaux Universitaires de Geneve, Geneva, Switzerland
- United Kingdom (19):
  - Royal Aberdeen Children's Hospital, Aberdeen
  - Royal Belfast Hospital for Sick Children, Belfast
  - Birmingham Children's Hospital, Birmingham
  - Bristol Royal Hospital for Children, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Noah's Ark Children's Hospital for Wales, Cardiff
  - Royal Hospital for Children, Edinburgh
  - Royal Hospital for Children, Glasgow
  - Leeds General Infirmary, Leeds
  - Leicester Royal Infirmary, Leicester
  - Alder Hey Children's Hospital, Liverpool
  - Great Ormond Street Hospital, London
  - Royal Manchester Children's Hospital, Manchester
  - Great North Children's Hospital, Newcastle upon Tyne
  - Nottingham Children's Hospital, Nottingham
  - Oxford Children's Hospital, Oxford
  - Sheffield Children's Hospital, Sheffield
  - University Hospital Southampton, Southampton
  - The Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: No